CLINICAL TRIAL: NCT02337504
Title: Developing and Assessing a Community Based Model of Antiretroviral Care
Acronym: ARTCo-ops
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moi University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, ABRAHAM M. SIIKA, MBChB, MMed, MS, Professor, Moi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GH000765
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: HIV
MeSH Terms: interventions — Delivery of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clinic-based care (No Intervention): Will receive HIV care at the clinic from the nurses and clinical officer on their regular schedule
- Community-based care (Active Comparator): Will receive HIV care in their community from a community health worker every month as part of a group of 6-10 people
  Interventions: Other: community-based care

INTERVENTIONS:
Other: community-based care — Will receive HIV care in the community and not in the clinic which is the normal standard of care
  Arms: Community-based care

SUMMARY:
Tremendous efforts and resources have been expended by the global community to ensure that antiretroviral therapy (ART) is available and accessible to all that need it. Despite these, less than a half of Human Immunodeficiency Virus (HIV)-infected patients requiring ART in sub-Saharan Africa (SSA) are receiving it. Some of the most significant barriers to attaining universal access to ART in this region include large distances that patients have to travel to clinic, time spent in accessing care and a significant shortage of human resources. In order to address these challenges the World Health Organization (WHO) advocates alternative care models especially those that incorporate task-shifting to lower cadre health care workers and lay persons. Unfortunately, few such alternative care models have been identified and very little data exist on their long-term outcomes.

With this project we will develop and assess an alternative care model that is established on the platform of a HIV-infected peer-group (ART Co-op) and facilitated by community health workers (CHW's). This model of care is intended to decentralize ART services and bring them closer to the patients. Specifically, we will:

1. Develop an acceptable and sustainable model for extending HIV care and treatment into the community.
2. Perform a pilot study comparing the outcomes of patients enrolled in the ART Co-ops program to those receiving standard of care.
3. Determine the cost savings and cost effectiveness of ART Co-ops.

DETAILED DESCRIPTION:
Universal Access to ART: Since 2003 there has been a concerted international effort to increase access to ART for HIV-infected individuals living in low and middle income countries.[1-6] Despite the substantial increase in the number of people receiving ART in SSA, by the end of 2010 only 49% of the 10,400,000 persons in need of ART were receiving treatment.[7-8] This is far short of the universal ART access goal of ≥80% of those in need of treatment.[2] Given that SSA commands only 3% of the world's health care providers and contributes to only 1% of the global health care expenditures, a significant barrier to meeting this goal is the profound shortage of infrastructure resources, most specifically, trained medical personnel.[9-10] With regard to Kenya, WHO estimates that the country will only be able to provide 25% of the 240,000 physicians needed to serve the country's population by 2015.[11] New initiatives under consideration such as "Test and Treat", Option B+ (ART for all pregnant women with lifelong maintenance) and treatment of index partners within HIV-discordant relationships will further tax the already strained health care work force.[12-22] As such, unless new care models can be developed that require fewer health care provider resources while maintaining optimal patient outcomes, the goal of universal access is unachievable.

Retention in Care: The high program attrition rates in SSA make achieving universal access even more complex. A meta-analysis of HIV-care programs in resource-constrained settings estimated one and two-year attrition rates (defined as death or lost to follow up (LTFU)) to be 22.6% (range 7-45%) and 25% (11-32%), respectively.[23] Of these approximately 41% were confirmed dead and 59% were LTFU. Patients LTFU represent heterogeneous outcomes including death, in care elsewhere, and disengaged from care.[24] Patients disengaged from care are at high risk of morbidity, mortality and transmitting HIV.[25-29] Despite the desirability of providing outreach to all patients LTFU, the cost of such programs frequently comes at the expense of expanding ART access. Geographic accessibility (distance to clinic and transportation costs) and shortages in health care personnel (excessive clinic waiting times) are documented barriers to retention.[24-25,30-35] As such, the optimal ART care model in resource constrained settings should minimize LTFU through reductions in transport time and costs as well as reducing clinic waiting time.

Task Shifting: In response to the severe shortage of health care workers in SSA, WHO and other organizations have advocated task shifting to lower cadre health care workers and lay individuals, including persons living with HIV (PLWHIV), in order to maximize patients' access to ART.[36-39] Such strategies decrease physician resource requirements, allow for decentralized ART delivery, and improve patient retention.[26,40-50] Médecins Sans Frontières (MSF) has developed a model of care which allows PLWHIV to become active participants in their own care and the care of other community members.[49]They successfully formed Community ART Groups (CAGs) to facilitate ART distribution, promote adherence, provide social support and monitor clinical status. During monthly group meetings a CAG member was chosen to represent each group at the clinic where each member's status was discussed and the group's monthly ART supply was picked up. Retention was exceptionally high with 97.5% patients remaining in care for a median follow-up period of 12.9 months (range 8.5-14 months).

Cost Effectiveness: Site-level cost studies of HIV care services have shown that human resource costs are a major determination of treatment scale-up costs and, as such, support the recommendations for task-shifting.[51-53] Despite this, only a few cost and cost-effectiveness studies have assessed alternative ART-delivery models.[54-59]

Justification for study:

This study proposes to refine and test a HIV-care model which utilizes CHWs and PLWHIV participating in their own care. The traditional ART-care model requires that patients attend monthly to every 4 monthly clinic visits conducted by a physician, clinical officer (CO) or a nurse. This model utilizes significant health worker and patient time resources,patient monetary resources for travel,and is a care-model disconnected from the local community. This proposal shifts the paradigm from intensive clinic-based supervision of ART-delivery to monitoring by community-based cooperative groups(ART Co-ops). We believe this innovative model will:1)decrease the amount of healthcare worker resources required to provide HIV-care;2)decrease costs;3)improve retention in care;and 4)increase access to ART and 5) maintain the durability of a patients ART regimen with limited health encounters.Given that this model utilizes systems and stakeholders already present in the community we believe that it is scalable to other resource constrained environments.ART Co-ops would provide a logical gateway from the community to HIV-clinics for HIV-infected individuals identified during" Test and Treat"initiatives and a community-based health resource for all HIV infected individuals(i.e., index partners in a discordant relationship and pregnant women).

Intended/potential use of study findings:

By achieving the specific aims we anticipate that we will develop a model of HIV-care that will minimize the number of health care providers needed to deliver HIV care while maximizing patient outcomes including durability of ART regimen and engagement and retention in care.We anticipate that such a model will be scalable to other settings in SSA as the resources necessary for this model exist in most communities within the region. Adoption of such models has the potential to allow for more cost effective delivery of ART-care in resource-constrained settings.

Study design/locations:

We will conduct formative research (assessment of secondary data, FGDs and KIIs) to guide the development and refinement of the ART Co-ops model as proposed in Specific Aim 1. A randomized prospective trial will compare the outcomes of subjects enrolled in the ART Co-ops Model to those receiving standard of care in Specific Aim 3. This study will be conducted at the AMPATH Partnership clinic in Kitale, Kenya, part of an HIV care and treatment program currently operating in 108 clinics in western Kenya [60-61]. The AMPATH clinic in Kitale currently has over 19,000 patients enrolled with >12,000 on ART. This is one of AMPATHs most rapidly growing clinic populations which makes it an ideal site for studying and implementing the use of a community care model.

Objectives:

Our long term goal is the development and successful implementation of an HIV care system that can facilitate the achievement of universal access to and maximize retention in ART programs in SSA. The major objective of this proposal is to develop and assess a community-based ART delivery model established on the platform of a HIV-infected peer-group (ART Co-op) and facilitated by CHWs. Our central hypothesis is that the durability of the patient's ART regimen (requiring no change to second line for failure) will remain equivalent to those seen in clinic regularly and that clinic outcomes (such as adherence to visits (clinic visits for the control group and ART Co-ops for the intervention group), retention in care (receiving care or being seen in an ART Co-op group within 3 months of the last scheduled visit), adherence to ART(>90s% ART taken on time))will be similar between this community-based model and the standard of care. We base this hypothesis on our previous studies utilizing task-shifting to provide ART care as well as recent data from Mozambique[49]on the use of community ART-Groups.

Aims/Hypotheses:

SA1: Develop an acceptable model for extending HIV care and treatment into the community.

H1: Information gathered through FGDs and KIIs will allow refinements in the ART Co-op model that will promote community and patient acceptance.

SA2: Develop a sustainable model for extending HIV care and treatment into the community.

H2: ART Co-ops can be assembled and managed with the assistance of CHWs.

SA3: Perform a pilot study comparing the outcomes of patients enrolled in the ART Co-ops program to those receiving standard of care.

H3a: Adherence to HIV-care visits (Co-op group meetings and /or clinic visits) and retention in care will be better in the ART Co-ops group.

H3b: Adherence to ART will be equivalent between the groups. H3c: Durability of the ART regimen will be equivalent between the groups. H3d: Patient perceived quality of life will be better in the ART Co-op group participants.

SA4: Determine the cost savings and cost effectiveness of ART Co-ops. H4a: ART Co-ops will generate cost savings to patients as well as the HIV care program.

H4b: ART Co-ops will be more cost effective than the standard of care when viewed from the program perspective.

General approach: A variety of approaches are used in the Specific Aims and their respective hypotheses. Specific Aim 1 is qualitative, utilizing the information gathered from KIIs and FGDs to inform refinements in the ART Co-op model necessary to promote community and patient acceptance and to prove its' sustainability within the community. Specific Aim 2 is process oriented, allowing for the assembly of ART Co-ops. Specific Aim 3 is comparative, allowing for an assessment of the ART Co-op groups as compared to the standard of care in their anticipated ability to improve adherence to HIV-care visits and patient's perceived quality of life (QOL), while maintaining an equivalent level of adherence and durability of ART regimen. Specific Aim 4 is descriptive, evaluating the interventions cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected
2. ≥18 years old
3. Have a current cluster of differentiation 4 (CD4)count ≥200cells/µl
4. Have an undetectable VL
5. Are clinically stable on ART for ≥ 6 months
6. A resident of a sub-location within the AMPATH Kitale clinic catchment area
7. Are willing to consent to participate

Exclusion Criteria:

1. Pregnant
2. Active opportunistic infection (OI)
3. Unable to consent for study participation due to physical or mental incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ART durability | 48 weeks
  Durability of ART regimen (ART failure). This is defined as the need to change ART regimens based on clinical (new or recurrent WHO 3 or 4 event), immunologic (CD4 count< pre-ART; ≥50% CD4 decrease from peak; persistent CD4<100) or virologic failure (VL>10,000 copies/mL). Durability of the patient's ART regimen (requiring no change to second line for failure) will remain equivalent to those seen in clinic regularly.

SECONDARY OUTCOMES:
Retention in care | 48 weeks
  Retention between the two groups will be compared at 48 weeks.
HIV VL (copies/mL) | 48 weeks
  Plasma viral load changes at 48 weeks will be measured
Quality of life | 48 weeks
  Quality of life at 48 weeks will be measured using a questionnaire
stigma | 48 weeks
  Stigma levels at 48 weeks will be measured using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Abraham M Siika, MD,MMED,MS, Principal Investigator — Moi University